Title: Effect of scapula-focused treatment with additional motor control exercises on pain

and disability in patients with subacromial pain syndrome: A Randomized Controlled Trial

Trial registration number. ClinicalTrials.gov (NCT02695524)

**Date**: 15/08/2019

1

# **BACKGROUND**

Subacromial pain syndrome (SPS) is a shoulder pain condition in which individuals report pain or discomfort associated with excessive overhead movements.<sup>1,2</sup> It corresponds to 44%-65% of all shoulder pain complaints<sup>2,3</sup> resulting in increased disability and reduced quality of life.<sup>4</sup> Factors associated with SPS include: disorders of scapula and clavicle kinematics,<sup>5</sup> glenohumeral stiffness and instability,<sup>6</sup> muscle weakness or disorders in motor control.<sup>7</sup>

The scapula plays an important role in absorption and energy transfer to maximize levels of upper limb freedom.<sup>8</sup> Periscapular muscles act synergistically to allow scapulohumeral coupled movements. In the last decade scapula assessment and treatment focused on "motor control exercises" has become ubiquitous for the rehabilitation process of painful shoulder. The latest systematic review with meta-analysis on the on the efficacy of exercises demonstrated that interventions focused on the scapula should be considered in treating SPS, provide benefits with short-term results for shoulder pain, function<sup>9</sup> and abduction ROM.<sup>9,10</sup>

The studies included in the meta-analysis that observed the additional effects of motor control exercises or scapula stabilization present important methodological limitations such as the absence of concealed allocation, blind subjects, blind assessor and absence of intention-to-treat analysis<sup>11,12</sup> that contribute to the low quality of evidence. Therefore, there is a need for further research through high-quality RCT that adequately assess the effects of scapula motor control exercises on clinical outcomes.

#### **OBJECTIVE**

Determine the effect of adding scapular motor control exercises to a scapula-focused program on disability, pain, muscle strength, and ROM in patients with Subacromial Pain Syndrome.

# **DESIGN OVERVIEW**

Controlled, randomized, superiority clinical trial, prospectively registered, two-arms, parallel, blind assessor, blind patient, and allocation concealment. All methodological steps were described by Consolidated Stands of Reporting Trials (CONSORT).

# **METHODS**

## **Setting and Participants**

Individuals with SPS were recruited from March 2016 to June 2017 by the local health system. The trial was conducted in an outpatient physical treatment service provided by the local health system. This study was approved by the University Research Ethics Committee (CAAE:52563216.0.0000.5414). All participants were informed about the procedures and signed the consent form.

**Inclusion Criteria:** participants with a history of shoulder pain for more than one week, located in the shoulder anterior-proximal region, with positive results for 3 out of 5 SPS tests:

1) Neer; 2) Hawkins-Kennedy; 3) painful arc; 4) pain or weakness resistant to external rotation, and 5) Jobe.<sup>13</sup>

**Exclusion criteria:** history of shoulder trauma or surgery; total rotator cuff or biceps brachii tendon rupture (imaging exam or self-report); practitioners of sports activities involving the

upper limbs; individuals with neurological disorders and alterations in cognitive function (e.g. stroke, epilepsy, multiple sclerosis, Parkinson's disease and peripheral neuropathy); shoulder pain for of primary involvement in the cervical or thoracic region; systemic disease involving the joints (e.g. rheumatoid arthritis); carpal tunnel syndrome; and those who underwent physiotherapeutic treatment of the shoulder in the last six months.

#### **Randomization and Intervention**

Simple randomization was carried out using a computer-generated schedule in Microsoft Excel (Microsoft Corporation, Redmond, Washington). Allocations were sealed, sequentially numbered envelopes, prepared by an individual not involved in the recruiting, assessment or treatment of the patients, and kept in a central locked location.

The envelopes were opened on the first day of the treatment, and the participants were randomly allocated into two treatment groups: the scapula-focused group (SFG) and the scapula motor control group (MCG). The subjects were treated individually and blinded regarding treatment allocation. Due to the nature of the interventions, it was not possible to blind the physical therapists that conducted the interventions.

The exercises for each group were based in a previously proposed protocol<sup>14</sup>. The patients assigned to the SFG performed 6 exercises with a focus on the periscapular muscles: 1) side lying external rotation with abduction at 0°15,16; 2) prone horizontal abduction with external rotation from 90° to 135°17,18; 3) Scapular punch<sup>19</sup>; 4) Knee Push<sup>20</sup>; 5) Full Can<sup>17,20</sup>; 6) Diagonal D1<sup>17</sup>. The exercise load was 60% of the one-repetition maximum (1-RM) during the first week because it was their first exposure to the exercises.<sup>21</sup> The weekly load progression averaged about 2.5% increase/wk up to -80% of 1-RM, according to the strength of each participant<sup>21</sup>. The exercises were performed in 3 series of 10 repetitions, with a 1-minute interval between repetitions during the first and fourth week.

From the fourth week on, the exercises were increased to 12 repetitions, and from the fifth to eighth week, to 15 repetitions.<sup>21</sup> The Push up plus<sup>17,22</sup> exercise with the feet flat on the floor was considered the progression exercise of the knee push.<sup>20</sup> The load progression for the push-up plus exercise takes place by lifting the feet on supports and could reach a height of 47.5 cm<sup>23</sup>.

The patients allocated to the MCG performed the scapula-focused exercises with the same progression, and six motor control exercises were added to this group. For this study, Motor control exercises were defined as retraction and depression movements of the scapula without external load (e.g., dumbbells and an elastic band) and associated with visual, verbal and kinestetic feedback in maintaining the posture. The six motor control exercises were always performed at the beginning of each session: A) Towel Slide<sup>24</sup>; B) Scapular Clock<sup>24</sup>; C) PNF Scapular<sup>24</sup>; D) Modified Inferior Glide<sup>25,26</sup>; E) Scapular Orientation Exercise (SOE)<sup>27,28</sup>; F) Protraction and retraction in front of a mirror. From the first to the third week, three series of 10 movements were performed for each exercise with verbal, visual, and kinesthetic feedback. On the fourth week, the exercises were increased to 12 movements, and visual feedback was removed. From the fifth to the eighth week, the exercises progressed to 15 repetitions, while verbal feedback was carried out only by the therapist. In both groups, the series of exercises were randomized into blocks at the beginning of each week.

## **Outcomes measures and Follow-up**

Shoulder function was considered the primary outcome; pain, treatment effect perception, satisfaction, kinesiophobia, strength, ROM, and scapula position were all considered the secondary outcomes.

**Function and pain:** The Brazilian version of Shoulder Pain and Disability Index (SPADI-Br) is valid and reliable for assessment of individuals with shoulder disorders<sup>29</sup> The Minimally Important Difference (MID) considered for the questionnaire was 10 points.<sup>30</sup> Higher scores indicated the worse condition.

A verbal, numerical pain rating scale was applied to measure the intensity of the pain. The values range from zero to ten and must be answered based on the pain intensity at the time of the test.<sup>31,32</sup>

**Treatment effect perception, satisfaction, and kinesiophobia**: The global perceived effect scale assessed patient perceptions of the effect of the treatment. For the assessment of patient satisfaction, The MedRisk<sup>34</sup> questionnaire was used. For assessment of the kinesiophobia level, the Tampa Scale of Kinesiophobia was applied.

Strength, ROM, and scapula position: Isometric strength assessment was carried out using a hand-held dynamometer (Lafayette<sup>®</sup>, Lafayette Instrument Company, Ind., USA). Muscle strength measurements were performed in abduction, adduction, internal and external arm rotation<sup>36</sup> and for specific muscles, of the serratus anterior, upper, middle and lower trapezius<sup>37</sup>.

For the ROM assessment, a digital inclinometer (Lafayette<sup>®</sup>, Lafayette Instrument Company, Ind., USA) was used during flexion, abduction and internal and external rotation active movements<sup>38</sup>. Upward rotation and scapula anterior/posterior tilt movements were also evaluated<sup>37,39,40</sup>.

### **STATISTICAL ANALYSES:**

**Sample size calculation:** Was performed with G\*Power 3.1 for Windows (Universität Kiel, Germany) based on the primary study outcome assessed by SPADI-Br questionnaire. The

sample was calculated based on the questionnaire's capacity to detect a 10-point difference in the global outcome score (SD=11.7), considering the clinically relevant difference, alpha 0.05, power 80% and considering a 20% sample loss.

Statistical analysis: Statistical analysis followed the intention-to-treat concept<sup>41,42</sup> using the Statistical Package for the Social Sciences Software (SPSS). The linear mixed-effect model was applied for the primary and secondary variables. In the model, "Time" and "group" were considered fixed effects, whereas the participants were considered the random effect. The time by group interaction was included in the analysis to assess the difference effect between the groups at each follow-up, and the dependent variable baseline value was included as a covariate for the correction of possible differences. The significance level was 0.05 for all analyses. The calculations of the effect size (ES) and Minimal Important Difference was carried out according to Armijo-Olivo et al<sup>43</sup>. The ES is calculated by dividing the difference between group mean scores by the pooled standard deviation of the 2 groups.

$$ES - \frac{X_{G1}-X_{G2}}{Spooled}$$
 and  $S_{pooled} - \frac{\sqrt{S_1^2(n1-1)+S_2^2(n2-1)}}{n1+n2-2}$ 

The effect size values were considered small (up to 0.2), moderate (0.5), and large (equal or above 0.8)<sup>44</sup>. Statistical analysis followed the intention-to-treat concept and was carried out by a researcher not involved in the evaluation and treatment protocols. The strength measures were examined with normalization to body weight (strength in kilograms/ kilogram of body weight X 100).

### References:

- Camargo PR, Haik MN, Ludewig PM, *et al.* Effects of strengthening and stretching exercises applied during working hours on pain and physical impairment in workers with subacromial impingement syndrome. *Physiother Theory Pract* 2009;25:463–75. doi:10.3109/09593980802662145
- 2 Michener LA, McClure PW, Karduna AR. Anatomical and biomechanical mechanisms of subacromial impingement syndrome. *Clin Biomech* 2003;18:369–79. doi:10.1016/S0268-0033(03)00047-0
- 3 Van Der Windt DAWM, Koes BW, Boeke AJP, *et al.* Shoulder disorders in general practice: Prognostic indicators of outcome. *Br J Gen Pract* 1996;46:519–23.
- 4 Chipchase LS, O'Connor DA, Costi JJ, *et al.* Shoulder impingement syndrome: Preoperative health status. *J Shoulder Elb Surg* 2000;9:12–5.
- Lawrence RL, Braman JP, Staker JL, *et al.* Comparison of 3-Dimensional Shoulder Complex Kinematics in Individuals With and Without Shoulder Pain, Part 2: Glenohumeral Joint. *J Orthop Sport Phys Ther* 2014;44:646-B3. doi:10.2519/jospt.2014.5556
- 6 Ludewig PM, Reynolds JF. The Association of Scapular Kinematics and Glenohumeral Joint Pathologies. *J Orthop Sport Phys Ther* 2009;39:90–104. doi:10.2519/jospt.2009.2808
- Phadke V, Camargo P, Ludewig P. Scapular and rotator cuff muscle activity during arm elevation: A review of normal function and alterations with shoulder impingement. *Rev Bras Fisioter* 2009;27:320–31. doi:10.1002/nbm.3066.Non-invasive
- McQuade KJ, Borstad J, de Oliveira AS. Critical and Theoretical Perspective on Scapular Stabilization: What Does It Really Mean, and Are We on the Right Track? *Phys Ther* 2016;96:1162–9. doi:10.2522/ptj.20140230
- 9 Saito H, Harrold ME, Cavalheri V, *et al.* Scapular focused interventions to improve shoulder pain and function in adults with subacromial pain: A systematic review and meta-analysis. *Physiother Theory Pract* 2018;3985:1–18. doi:10.1080/09593985.2018.1423656
- Bury J, West M, Chamorro-Moriana G, *et al.* Effectiveness of scapula-focused approaches in patients with rotator cuff related shoulder pain: A systematic review and meta-analysis. *Man Ther* 2016;25:35–42. doi:10.1016/j.math.2016.05.337
- Başkurt Z, Başkurt F, Gelecek N, *et al.* The effectiveness of scapular stabilization exercise in the patients with subacromial impingement syndrome. *J Back Musculoskelet Rehabil* 2011;24:173–9. doi:10.3233/BMR-2011-0291
- Shah M, Sutaria J, Khant A. Effectiveness of Scapular Stability Exercises in the Patient With the Shoulder Impingement Syndrome. *Indian J Phys Ther 2014;2(1)79-84* 2014;2:79–84.
- 13 Michener LA, Walsworth MK, Doukas WC, *et al.* Reliability and diagnostic accuracy of 5 physical examination tests and combination of tests for subacromial impingement. *Arch Phys*

- Med Rehabil 2009;90:1898-903. doi:10.1016/j.apmr.2009.05.015
- Hotta GH, Santos AL, McQuade KJ, et al. Scapular-focused exercise treatment protocol for shoulder impingement symptoms: Three-dimensional scapular kinematics analysis. Clin Biomech Published Online First: 2017. doi:10.1016/j.clinbiomech.2017.12.005
- De Mey K, Danneels L, Cagnie B, *et al.* Conscious Correction of Scapular Orientation in Overhead Athletes Performing Selected Shoulder Rehabilitation Exercises: The Effect on Trapezius Muscle Activation Measured by Surface Electromyography. *J Orthop Sport Phys Ther* 2013;43:3–10. doi:10.2519/jospt.2013.4283
- Hess SA, Richardson C, Darnell R, *et al.* Timing of Rotator Cuff Activation During Shoulder External Rotation in Throwers With and Without Symptoms of Pain. *J Orthop Sport Phys Ther* 2005;35:812–20. doi:10.2519/jospt.2005.35.12.812
- Escamilla RF, Yamashiro K, Paulos L, *et al.* Shoulder muscle activity and function in common shoulder rehabilitation exercises. *Sports Med* 2009;39:663–85. doi:10.2165/00007256-200939080-00004
- De Mey K, Cagnie B, Van De Velde A, *et al.* Trapezius Muscle Timing During Selected Shoulder Rehabilitation Exercises. *J Orthop Sport Phys Ther* 2009;39:743–52. doi:10.2519/jospt.2009.3089
- Reinold MM, Escamilla R, Wilk KE. Current Concepts in the Scientific and Clinical Rationale Behind Exercises for Glenohumeral and Scapulothoracic Musculature. *J Orthop Sport Phys Ther* 2009;39:105–17. doi:10.2519/jospt.2009.2835
- Maenhout A, Van Praet K, Pizzi L, *et al.* Electromyographic analysis of knee push up plus variations: what is the influence of the kinetic chain on scapular muscle activity? *Br J Sports Med* 2010;44:1010–5. doi:10.1136/bjsm.2009.062810
- American College of Sports Medicine position stand. Progression models in resistance training for healthy adults. *Med Sci Sports Exerc* 2009;41:687–708. doi:10.1249/MSS.0b013e3181915670
- Weiser WM, Lee TQ, McMaster WC, *et al.* Effects of simulated scapular protraction on anterior glenohumeral stability. *Am J Sports Med* 1999;27:801–5.
- Lear LJ, Gross MT. An electromyographical analysis of the scapular stabilizing synergists during a push-up progression. *J Orthop Sports Phys Ther* 1998;28:146–57. doi:10.2519/jospt.1998.28.3.146
- Voight ML, Thomson BC. The Role of the Scapula in the Rehabilitation of Shoulder Injuries. *J Athl Train* 2000;35:364–72. doi:10.1016/B978-044306701-3.50053-0
- Ben Kibler W, Sciascia AD, Uhl TL, *et al.* Electromyographic analysis of specific exercises for scapular control in early phases of shoulder rehabilitation. *Am J Sports Med* 2008;36:1789–98. doi:10.1177/0363546508316281
- 26 Ekstrom RA, Donatelli RA, Soderberg GL. Surface Electromyographic Analysis of Exercises

- for the Trapezius and Serratus Anterior Muscles. *J Orthop Sport Phys Ther* 2003;33:247–58. doi:10.2519/jospt.2003.33.5.247
- 27 Mottram SL, Woledge RC, Morrissey D. Motion analysis study of a scapular orientation exercise and subjects' ability to learn the exercise. *Man Ther* 2009;14:13–8. doi:10.1016/j.math.2007.07.008
- 28 Mottram S. Dynamic stability of the scapula. *Man Ther* 1997;2:123–31. doi:https://doi.org/10.1054/math.1997.0292
- Martins J, Napoles B V., Hoffman CB, *et al.* The Brazilian version of Shoulder Pain and Disability Index: translation, cultural adaptation and reliability. *Brazilian J Phys Ther* 2010;14:527–36. doi:10.1590/S1413-35552010000600012
- 30 Roy JS, Macdermid JC, Woodhouse LJ. Measuring shoulder function: A systematic review of four questionnaires. *Arthritis Care Res* 2009;61:623–32. doi:10.1002/art.24396
- Farrar JT, Young JP, LaMoreaux L, *et al.* Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. *Pain* 2001;94:149–58.
- Turk DC, Dworkin RH, Allen RR, *et al.* Core outcome domains for chronic pain clinical trials: IMMPACT recommendations. 2003;:337–345. doi:doi:10.1016/j.pain.2003.08.001
- Costa LOP, Maher CG, Latimer J, *et al.* Clinimetric testing of three self-report outcome measures for low back pain patients in Brazil: which one is the best? *Spine (Phila Pa 1976)* 2008;33:2459–63. doi:10.1097/BRS.0b013e3181849dbe
- de Fátima Costa Oliveira N, Oliveira Pena Costa L, Nelson R, *et al.* Measurement properties of the Brazilian Portuguese version of the MedRisk instrument for measuring patient satisfaction with physical therapy care. *J Orthop Sports Phys Ther* 2014;44:879–89. doi:10.2519/jospt.2014.5150
- de Souza FS, Marinho C da S, Siqueira FB, *et al.* Psychometric testing confirms that the Brazilian-Portuguese adaptations, the original versions of the Fear-Avoidance Beliefs Questionnaire, and the Tampa Scale of Kinesiophobia have similar measurement properties. *Spine (Phila Pa 1976)* 2008;33:1028–33. doi:10.1097/BRS.0b013e31816c8329
- Beshay N, Lam PH, Murrell GAC. Assessing the reliability of shoulder strength measurement: hand-held versus fixed dynamometry. *Shoulder Elb* 2011;3:244–51. doi:10.1111/j.1758-5740.2011.00137.x
- Cools AM, Johansson FR, Cambier DC, *et al.* Descriptive profile of scapulothoracic position, strength and flexibility variables in adolescent elite tennis players. *Br J Sports Med* 2010;44:678–84. doi:10.1136/bjsm.2009.070128
- Mullaney MJ, McHugh MP, Johnson CP, et al. Reliability of shoulder range of motion comparing a goniometer to a digital level. *Physiother Theory Pract* 2010;26:327–33. doi:10.3109/09593980903094230
- 39 Watson L. Balster SM, Finch C. et al. Measurement of scapula upward rotation: a reliable

- clinical procedure. Br J Sports Med 2005;39:599-603. doi:10.1136/bjsm.2004.013243
- 40 Scibek JS, Carcia CR. VALIDATION OF A NEW METHOD FOR ASSESSING SCAPULAR ANTERIOR-POSTERIOR TILT. *Int J Sports Phys Ther* 2014;9:644–56.
- Morden JP, Lambert PC, Latimer N, *et al.* Assessing methods for dealing with treatment switching in randomised controlled trials: A simulation study. *BMC Med Res Methodol* 2011;11:4. doi:10.1186/1471-2288-11-4
- 42 Elkins MR, Moseley AM. Intention-to-treat analysis. *J Physiother* 2015;61:165–7. doi:10.1016/j.jphys.2015.05.013
- Armijo-Olivo S, Warren S, Fuentes J, *et al.* Clinical relevance vs. statistical significance: Using neck outcomes in patients with temporomandibular disorders as an example. *Man Ther* 2011;16:563–72. doi:10.1016/j.math.2011.05.006
- Cohen J. Statistical Power Analysis for the Behavioral Sciences. 2nd ed. New York: : Lawrence Erlbaum Associates 1988.